CLINICAL TRIAL: NCT03934619
Title: Dolores One: Maximizing Functional Communication for Adults Using Non-Invasive Ventilation in the Acute Care Setting
Brief Title: Dolores One: Maximizing Functional Communication for Adults
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: change in clinical practice that led to ability to recruit subjects
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Chris Wells, EBP & Research Coordinator, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HP-00078386
Record Dates: First submitted 2019-04-15; First posted 2019-05-02 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Communication
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: This study will be a prospective study using a convenient cohort of 55 adult patients, who was using NIV, to pilot the effectiveness of the Dolores One to improve verbal communication. There will be no randomization and no control group. The design is a pretest / posttest mixed method in which the Easy of Communication Scale and the Intelligibility section of the Frenchay Dysarthria Assessment will be administered at base line and repeated once the Dolores One has been set up on the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Convenient cohort, non-randomized group will be enrolled to examine the effects of the Dolores One on improving the ease of communication and intelligibility
  Interventions: Device: Dolores One

INTERVENTIONS:
Device: Dolores One — Dolores One, which is a will be applied personal sounds amplification device, will be used to determine if it improves the ability to communication and improves intelligibility

SUMMARY:
Difficulties with communication for patients requiring mechanical ventilation is known to be a source of distress in the acute care setting. The inability to speak has been associated with increased psychological distress and increased feelings of fear and anger and impact negatively on patient participation with caregivers and their overall recovery. Developing and maintaining communication between patients and hospital staff reduces patient stress and increases patient satisfaction and part of the standard pf care. According to the new and revised The Joint Commission standards, hospitals must identify and document patients' communication needs and communicate with patients during their care in a manner that meets those needs. Using the Dolores One device for patients can improve the ease and efficiency of communication while they are in the acute care setting.

For non-speaking patients, nonverbal communication means are often used, including mouthing words and head nods to indicate yes/no responses. However, relying completely on nonverbal means can limit patient responses and lead to ineffective and frustrating communication exchanges. There have been several studies reviewing the negative effects of the inability to speak for intubated, mechanically ventilated patients. However, there is a need for more research to address communication difficulties in other mechanically ventilated populations, including patients receiving non-invasive ventilation and ventilator dependent tracheostomy patients.

The Dolores One is comprised of an acoustic throat sensor and positioned at the patient's neck with a soft adjustable collar. The sensor gathers vocal cord vibrations and transmits signals to a control unit, processes the sensor signal, and finally, generates the patient's voice. The smart signal processing automatically accommodates both weak forced voices and whispers, producing a voice output to allow for normal conversation in a patient's natural voice, free from the sounds of rushing air or equipment noises secondary to Non-Invasive Mechanical Ventilation (NIMV) systems.

The purpose of the study is to determine if the Dolores One devices can be used in the clinical acute care setting with patients in NIMV to improve their ability to communication as measured as ease to communicate and intelligibility, with family and the members of the medical team.

DETAILED DESCRIPTION:
Primary Aims:

1. Is to determine if the Dolores One device can significantly improve the ease of communication as measured by the Ease of Communication
2. Is to determine if the Dolores One device can significantly improve the intelligibility of communication as measured by the Intelligibility section of the Frenchay Dysarthria Assessment (FDA).

Design:

This study will be a prospective study using a convenient cohort of 55 adult patients, who was using NIMV, to pilot the effectiveness of the Dolores One to improve verbal communication. There will be no randomization and no control group. The design is a pretest / posttest mixed method in which the Easy of Communication Scale and the Intelligibility section of the FDA will be administered at base line and repeated once the Dolores One has been set up on the patient.

Methodology:

The respiratory therapists who are working in the Medical Intensive Care Unit (MICU) and 10 West will complete the initial screening for potential subjects based upon the study's eligibility criteria. The floor respiratory therapist will notify the Principle Investigator (PI) of a potential subject. The PI will either verify that the patient meets the eligibility criteria or will contact another member of the study team to verify eligibility, medically appropriateness to participate and consent the patient. To screen for medical appropriateness and minimize risk a member of the study team will have a conversation with medical team to determine medical stability as defined as patient having stable vitals on NIMV as defined by medical team parameters and nursing orders for the individual patient and on stable NIMV setting for 30 to 90 minutes as per respiratory therapy guidelines.

Once the consent has been obtained, the Speech Language Pathologist (SLP) will be notified and will obtain the data regarding the parameters of the NIMV and document current vital signs, which is standard practice for patient safety. Then the speech therapist will complete the baseline communication assessment using the Ease of Communication Scale and the Intelligibility section of the FDA. The Ease of Communication Scale is a self report 10 item questionnaire in which the subject rates their ability to communication while on NIMV. It is on a 5 item Likert scale and a total sum is recorded. For the Intelligibility Section of the FDA, the speech therapist will use a random table to select 5 short sentences or phrase in which there is a key word. The speech therapist will ask the subject to speak these phrase out loud. A volunteer staff member, who is unfamiliar with the list of possible sentences provided in the FDA, will be asked to write down the sentences the subject speaks. The SLP will score the intelligibility as a yes no response based upon the accuracy of the key word. Intelligibility will be reported as a percentage of correct responses. The statements will be randomized to decrease familiarity as well as there are over 140 nurses and 15 nurse aides and other various staff that work on these units that the speech therapist may obtain to as a volunteer. The volunteer pool is sufficient to decrease the likelihood of the volunteer being familiar with the statements to bias the test results. If a staff member who is assigned for daily care for this subject is unavailable, or unable to volunteer at time of testing, the Speech therapist will ask another staff member of the unit who has been educated regarding the study, to assist.

After preliminary data collection has been completed, the SLP will place the Dolores One on the patient and adjust sensor position and device volume to achieve optimal voice output. The SLP will position the Dolores One on either side of the neck to assure comfort and effective sound. It will not be applied to any area of skin rash or lesion. The device can be removed at any time and reapplied when the patient would like to speak. The Dolores One will be left with the patient to have the opportunity to use the device to communicate with their health care team and visitors for the next 24 to 36 hours. The speech therapist training session will take approximately 10 minutes to train the subject on the use and to practice prior to the therapist leaving.

The SLP will return between 24 and 36 hours from initial data collection, verify medical and NIMV stability, record vitals, obtain NIMV parameters, and repeat the Ease of Communication Scale and the Intelligibility Section of the FDA. After testing, this concludes the subjects participation in the study.

Other data that will be collected include, age, race, gender, unit location, NIMV Manufacture brand, NIMV setting: Fraction of Oxygen (FiO2), Positive End Expiratory Pressures (PEEP), inspiratory pressure, minute ventilation, and patient vitals (heart rate, blood pressure, respiratory rate and oxygen saturation), leak percentage , and primary diagnosis. This data will be collected at the time pre and post application of the Dolores One prior to completing the Ease of Communication Survey and the Intelligibility Section of FDA.

Prior to the start of this study the unit will receive education regarding the study and the general use of the Dolores One. Providers will be notified by providing educational materials in the team report rooms and will notify the attending as well as the medical director for the units

Separate training regarding the study, use of the Dolores One and screening criteria will be given to the respiratory therapy department via their hand off meetings. This has been approved by respiratory leadership. The Respiratory Therapist (RT) will be provided with the eligibility criteria to improve screening process.

ELIGIBILITY:
Inclusion Criteria:

* Requires NIMV
* Uses a full face mask
* Using a University of Maryland Medical Center (UMMC) device
* Medically stable as determined by the medical team (register nurse (RN) and licensed independent provider)
* The patient is stable on NIMV which measure same settings for a period 30 to 90 minutes as per RT guidelines
* Glasgow Coma Scale (GCS) 15
* Subjects speak English
* Skin is intact in the area where the Dolores One would be placed.

Exclusion Criteria:

* Patient is unable to consent self for the study
* Pre-existing speech, language, voice or cognitive deficits
* NIMV setting that exceeds the following prescription: FIO2 > .60; Peep > 12 mmHg, inspiratory pressure > 15 mmHg

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Change in the Easy of Communication Scale | Testing is at baseline, and 24-36 hours after use of the Dolores One
  Easy of Communication Scale is a self reported 10 item questionnaire where the subjects rate their perception of the ease to communicate. It is scored on a 5 point likert scale (0 to 4) with a range of 0-40. The investigators are examining the change in communication without and with the use of the Dolores One device. The higher the score the more difficulty the subject perceives it is to communicate with other.
Change in the Intelligibility Subscale of the Frenchay Dysarthria Assessment Tool | Testing is at baseline and 24 to 36 hours after use of the Dolores One
  The Intelligibility Score is a subscale of the Frenchay Dysarthria Assessment Tool that examines motor speech deficits. The Intelligibility Subscales examines the precision of articulation. This subscale involves the subject speaking 5 randomized short phrases and the intelligibility is scored as a yes / no based upon accuracy of a volunteer repeating the phrase accurately. The subscale has a range of 0-5 with 5 being normal and has a minimally detectable change of 1 being significant.

CONTACTS AND LOCATIONS:
Overall Officials: Chris L Wells, PhD, PT, Principal Investigator — Univeristy of Maryland Baltimore
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Professional Presentations and possible manuscript
Supporting Information: Study Protocol, SAP
Time Frame: 2 years
Access Criteria: Professional Speech conference; possibly respiratory therapy conference. Will also be shared within our organization as it relates to use of the device is we have positive findings

REFERENCES:
- [Background] Happ MB, Garrett K, Thomas DD, Tate J, George E, Houze M, Radtke J, Sereika S. Nurse-patient communication interactions in the intensive care unit. Am J Crit Care. 2011 Mar;20(2):e28-40. doi: 10.4037/ajcc2011433. PMID 21362711
- [Background] Khalaila R, Zbidat W, Anwar K, Bayya A, Linton DM, Sviri S. Communication difficulties and psychoemotional distress in patients receiving mechanical ventilation. Am J Crit Care. 2011 Nov;20(6):470-9. doi: 10.4037/ajcc2011989. PMID 22045144
- [Background] Magnus VS, Turkington L. Communication interaction in ICU--Patient and staff experiences and perceptions. Intensive Crit Care Nurs. 2006 Jun;22(3):167-80. doi: 10.1016/j.iccn.2005.09.009. Epub 2005 Nov 17. PMID 16298132
- [Background] Patak L, Wilson-Stronks A, Costello J, Kleinpell RM, Henneman EA, Person C, Happ MB. Improving patient-provider communication: a call to action. J Nurs Adm. 2009 Sep;39(9):372-6. doi: 10.1097/NNA.0b013e3181b414ca. No abstract available. PMID 19745632